CLINICAL TRIAL: NCT00654069
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter, Repeat-dose Study of the Safety and Efficacy of Acuroc Tablets Following Bunionectomy Surgery in Adult Patients
Brief Title: Safety/Efficacy Study of Oxycodone HCl/Niacin to Treat Pain After Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acura Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-ADF-105
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2008-04

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone; Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Tablet
  Interventions: Drug: Placebo
- Acurox 5/30mg (Active Comparator): Oxycodone HCl 5mg/Niacin 30mg tablet
  Interventions: Drug: Acurox 5/30 mg
- Acurox 7.5/30 (Placebo Comparator): Oxycodone HCl 7.5mg/Niacin 30mg tablet
  Interventions: Drug: Acurox 7.5/30

INTERVENTIONS:
Drug: Placebo — 2 tablets every 6 hours for 48 hours
  Other Names: Placebo Tablet
  Arms: Placebo
Drug: Acurox 5/30 mg — 2 tablets every 6 hours for 48 hours
  Other Names: oxycodone/niacin 5/30mg
  Arms: Acurox 5/30mg
Drug: Acurox 7.5/30 — 2 tablets every 6 hours for 48 hours
  Other Names: oxycodone/niacin 7.5/30mg
  Arms: Acurox 7.5/30

SUMMARY:
The purpose of this study is to determine whether oxycodone HCl and niacin are effective in the treatment of pain following bunionectomy surgery.

DETAILED DESCRIPTION:
This was a Phase III, randomized, double blind, placebo controlled, multicenter, repeat dose study of the safety and efficacy of 2 dose levels of Acurox™ Tablets versus placebo for the treatment of moderate to severe postoperative pain following bunionectomy surgery.

Patients underwent a primary unilateral first metatarsal bunionectomy with or without ipsilateral hammer toe repair during standardized local anesthesia with intravenous (IV) sedation. Eligible patients who reported moderate or severe pain within 6 hours after surgery entered the Treatment Phase and were randomized to 1 of 3 double blind treatments: placebo tablets or 1 of 2 dose levels of Acurox™ Tablets (ocyxcodone HCl/niacin). The Treatment Phase continued with study medication every 6 hours (irrespective of rescue medication use) for 48 hours (8 doses of study medication). Toradol (ketorolac tromethamine) was available as a rescue medication upon request.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female at least 18 years of age
* For women of child-bearing potential: woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Patient is scheduled to have a bunionectomy
* Patient must be willing to stay at the study site for at least 48 hours from the initial dose of study medication post-surgery

Exclusion Criteria:

* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen
* Patient is hypersensitive to any of the medications to be used in the study
* Patient has taken another investigational drug within 30 days prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

REFERENCES:
- [Derived] Daniels SE, Spivey RJ, Singla S, Golf M, Clark FJ. Efficacy and safety of oxycodone HCl/niacin tablets for the treatment of moderate-to-severe postoperative pain following bunionectomy surgery. Curr Med Res Opin. 2011 Mar;27(3):593-603. doi: 10.1185/03007995.2010.548291. Epub 2011 Jan 13. PMID 21231862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 405 post-bunionectomy patients
Pre-assignment Details: Subjects dose immediately post-surgery when pain intensity was equal to or greater than moderate. Dosed and followed for 48 hours.
Groups:
- Placebo: 2 Tablets Every 6 Hours
- Acurox 5/30mg: 2x oxycodone 5mg/naicin 30mg every 6 hours
- Acurox 7.5/30mg: 2x oxycodone 7.5mg/naicin 30mg every 6 hours
Period: Overall Study
Arm/Group | Placebo | Acurox 5/30mg | Acurox 7.5/30mg
Started | 136 | 135 | 134
Completed | 119 | 124 | 116
Not Completed | 17 | 11 | 18

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 2x Placebo Tablets
- Acurox 5/30: 2x oxycodone/niacin 5/30mg tablets
- Acurox 7.5/30: 2x oxycodone/niacin 7.5/30mg tablets
- Total: Total of all reporting groups
Arm/Group | Placebo | Acurox 5/30 | Acurox 7.5/30 | Total
Number analyzed (Participants) | 136 | 135 | 134 | 405
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 117 | 117 | 116 | 350
  >=65 years | 19 | 18 | 18 | 55
Age, Continuous [Mean (Full Range); unit: years] | 42.0 [18 to 71] | 41.8 [18 to 76] | 41.6 [18 to 77] | 41.8 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 125 | 120 | 359
  Male | 22 | 10 | 14 | 46
Region of Enrollment [Number; unit: participants]
  United States | 136 | 135 | 134 | 405

OUTCOME MEASURES:

1. Primary Outcome: SPID48
Description: Time weighted Sum of Pain Intensity Differences over the first 48 hours (SPID48) is the sum of the Pain Intensity Difference (PID) scores observed at 0.5 , 1, 2, 3, 4, 5, 6, 12, 18, 24, 30, 36, 42, and 48 hours post-dose. Pain Intensity scores at each timepoint are based on a 100 mm visual analog scale (VAS) from 0 = no pain to 100 = worst pain imaginable. PID is calculated as the timepoint score less the baseline pre-dose score (i.e. PID.5 = PI.5 - PI0).
  SPID48 = the PID for each timepoint multiplied by a time weighting factor; which is the difference (in hours) between the PID observation and prior observation. SPID48 = PID.5*.5 + PID1*.5 + PID2*1 + PID3*1 + PID4*1 + PID6*2 +PID12*6 + PID18*6 +PID24*6 + PID30*6 + PID36*6 + PID42*6 + PID48*6. The maximum SPID48 value is 4,800 (assumes PI0 of 100 and a PI of 0 at all subsequent timepoints) with a midpoint SPID48 of 2,400 (PI0=50 and PI of 0 at all subsequent readings).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo Tablet
- Acurox 5/30: oxycodone 5mg/niacin 30mg
- Acurox 7.5/30: oxycodone 7.5mg/niacin 30mg
Arm/Group | Placebo | Acurox 5/30 | Acurox 7.5/30
Number analyzed (Participants) | 119 | 124 | 116
score on a scale | 604.48 (1124.857) | 998.46 (1102.164) | 1224.97 (1128.569)

ADVERSE EVENTS:
Time Frame: 48 hours
Groups:
- Placebo: Placebo Pill
Arm/Group | Placebo | Acurox 5/30 | Acurox 7.5/30
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/135 | 0/134
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/135 | 0/134
Other Adverse Events (participants affected / at risk) | 51/136 | 104/135 | 117/134
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=136) | Acurox 5/30 (N=135) | Acurox 7.5/30 (N=134)
Nausea (Gastrointestinal disorders) | 23 (23) | 68 (68) | 83 (83)
Vomiting (Gastrointestinal disorders) | 14 (14) | 46 (46) | 67 (67)
Dizziness (Nervous system disorders) | 6 (6) | 22 (22) | 32 (32)
Headache (Nervous system disorders) | 3 (3) | 13 (13) | 11 (11)
Somnolence (Nervous system disorders) | 2 (2) | 8 (8) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 17 (17) | 13 (13)
Flushing (Vascular disorders) | 2 (2) | 22 (22) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No